CLINICAL TRIAL: NCT03048110
Title: A Phase I, Non-randomized, Open-label, Fixed-sequence Study to Investigate the Effect of a Probe CYP3A4 Inhibitor and Inducer on the Pharmacokinetics of BAY1841788 (ODM 201) in Healthy Male Volunteers
Brief Title: Drug-drug Interaction (DDI) Study to Assess ODM-201 as a Victim of CYP3A4 Inhibition or Induction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17726; 2016-004469-20 (EudraCT Number)
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Biological Availability
MeSH Terms: interventions — darolutamide; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ODM-201 (Experimental): All subjects will receive a single dose of BAY1841788 (ODM-201) (600 mg) in the first treatment period of the study, then all subjects will receive twice daily 200 mg itraconazole on 1 day and once daily 200 mg itraconazole for the following 6 days and a single dose of BAY1841788 (ODM-201) (600 mg) in the second treatment period, then all subjects will receive once a day 600 mg rifampicin for 10 days and a single dose of BAY1841788 (ODM-201) (600 mg) in the third treatment period
  Interventions: Drug: BAY1841788 (ODM-201); Drug: Itraconazole; Drug: Rifampicin

INTERVENTIONS:
Drug: BAY1841788 (ODM-201) — In Period 1, 600 mg single dose administered as 2x300 mg tablets on Study Day 1, In Period 2, 600 mg single dose administered as 2x300 mg tablets on Study Day 5, In Period 3, 600 mg single dose administered as 2x300 mg tablets at Study Day 8.
Drug: Itraconazole — 200 mg twice daily (BID) administered as 2 x 100 mg capsules per dose in treatment period 2 on Study Day 1, 200 mg once daily (QD) administered as 2 x 100 mg capsules per dose in treatment period 2 on Study Days 2 to 7.
Drug: Rifampicin — 600 mg QD administered as 1 x 600 mg tablet per dose in treatment period 3 on Study Days 1 to 10.

SUMMARY:
Evaluate the effect of a probe CYP3A4 inhibitor and inducer on the pharmacokinetics of BAY1841788 (ODM-201)

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject - as determined by the investigator or medically qualified designee based on medical evaluations including medical history, physical examination, laboratory tests and cardiac monitoring.
* Gender: Male.
* Age: 45 to 65 years (inclusive) at the screening visit.
* Race: White.
* Body mass index (BMI): ≥18.0 and ≤30 kg/m^2.
* Agree to use condoms as an effective contraception barrier method and refrain from sperm donation during the whole study (starting after informed consent) and for 3 months after the end of treatment with ODM-201. In addition, participants must agree to utilize a second reliable method of contraception simultaneously. The second method which has to be used by a female partner of childbearing potential can be one of the following methods: diaphragm or cervical cap with spermicide or intra-uterine device or hormone-based contraception.
* Results of alcohol tests are negative at screening and on Study Day -1.

Exclusion Criteria:

* Medical and surgical history
* Existing relevant diseases of vital organs (e.g. liver diseases, heart diseases), central nervous system (for example seizures) or other organs (e.g. diabetes mellitus).

Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.

* Febrile illness within 1 week before the first study drug administration.
* A medical history of risk factors for Torsades de Pointes (e.g. family history of Long QT Syndrome) or other arrhythmias.
* Known severe allergies, non-allergic drug reactions, or (multiple) drug allergies (excluding untreated, asymptomatic seasonal allergies like non-severe hay fever during the time of study conduct).
* Known history of hypersensitivity (or known allergic reaction) to itraconazole, rifampicin or ODM-201.
* Relevant hepatic disorders like cholestasis, disturbances of bilirubin metabolism, any progressive liver disease.
* Relevant renal disorders like recurrent glomerulonephritis, renal injury, and renal insufficiency. However, a history of a single episode of uncomplicated nephrolithiasis will not prevent participation.
* Subjects with porphyria.
* Subjects with diagnosed malignancy within the past 5 years except for cured skin basal carcinoma.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Time Zero to 72 Hours (AUC[0-72h]) of Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose to 72 hours post dose of darolutamide
  Area under the concentration versus time curve from time zero to 72 hours of Darolutamide after single dose administration in plasma were measured.
Maximum Observed Concentration (Cmax) of Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Maximum observed concentration after single dose administration in plasma were measured.
Area Under the Concentration Versus Time Curve From Time Zero to 72 Hours (AUC[0-72h]) of (S,R)-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Area under the concentration versus time curve from time zero to 72 hours of (S,R)-Darolutamide in plasma after single dose administration of Darolutamide were measured.
Maximum Observed Concentration (Cmax) of (S,R)-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Maximum observed concentration of (S,R)-darolutamide in plasma after single dose administration of darolutamide were measured.
Area Under the Concentration Versus Time Curve From Time Zero to 72 Hours (AUC[0-72h]) of (S,S)-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Area under the concentration versus time curve from time zero to 72 hours of (S,S)-darolutamide in plasma after single dose administration of darolutamide were measured.
Maximum Observed Concentration (Cmax) of (S,S)-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Maximum observed concentration of (S,S)-darolutamide in plasma after single dose administration of darolutamide were measured.
Area Under the Concentration Versus Time Curve From Time Zero to 72 Hours (AUC[0-72h]) of Keto-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Area under the concentration versus time curve from time zero to 72 hours (AUC[0-72h]) of keto-Darolutamide in plasma after single dose administration of darolutamide were measured.
Maximum Observed Concentration (Cmax) of Keto-Darolutamide in Plasma After Single Dose Administration of Darolutamide | Pre dose up to 72 hours post dose of darolutamide
  Maximum observed concentration of keto-darolutamide in plasma after single dose administration of darolutamide were measured.

SECONDARY OUTCOMES:
Number of Subjects With Study Drug-Related Treatment Emergent Adverse Events (TEAEs) | From start of study drug administration up to 30 days after last dose of study medication
  An adverse event (AE) was any untoward medical occurrence in subject who received study drug without regard to possibility of causal relationship. AEs that started or worsened after first administration of study medication up to 30 days after end of treatment with study medication were considered to be treatment-emergent (TE). AEs that occurred on study drug administration were termed as study drug related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany